CLINICAL TRIAL: NCT00539045
Title: Diagnostic Utility of Contrast Echocardiography for Detection of Left Ventricular Thrombi Post ST Elevation Myocardial Infarction
Brief Title: Diagnostic Utility of Contrast Echocardiography for Detection of LV Thrombi Post ST Elevation Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Lantheus Medical Imaging (Industry)
Responsible Party: Principal Investigator, Jonathan W. Weinsaft, Associate Professor, Weill Medical College of Cornell University
Other Study IDs: 0610008782
Record Dates: First submitted 2007-10-02; First posted 2007-10-03 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Thrombus; Myocardial Infarction
Keywords: myocardial infarction, thrombus
MeSH Terms: conditions — Thrombosis; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: The study population will consist of patients who are admitted to The New York Presbyterian Hospital-Weill Medical College of Cornell University (NYP-WMC) with ST elevation myocardial infarctions (STEMI). STEMI will be established based on standard clinical and ECG criteria.

SUMMARY:
This is a cross-sectional study of post myocardial infarction patients which is designed to determine the prevalence of left ventricular thrombi (blood clots) using non-contrast echocardiography and to compare this with the prevalence of left ventricular thrombi using contrast echocardiography. Secondary aims of this study are (1) to identify clinical and imaging correlates of left ventricular thrombi, and (2) to compare quantitative measurements of left ventricular chamber size, function, and myocardial mass using contrast and non-contrast echocardiography.

DETAILED DESCRIPTION:
People that experience heart attacks ("myocardial infarctions") are at increased risk for stroke, possibly due to formation of blood clots ("left ventricular thrombi"), which may break loose from the heart and travel to other organs. While echocardiography is a test commonly employed for thrombus detection, prior studies have yielded heterogeneous findings regarding prevalence and predictors. Echocardiographic contrast ("perflutren lipid microspheres") are FDA approved imaging agents that have been shown to improve thrombus detection in selected populations. However, the decision to use contrast is often predicated upon results of non-contrast echocardiography, a diagnostic strategy that hasn't been well studied. This study is designed to test whether echocardiographic contrast improves thrombus detection following myocardial infarction. Participants will undergo non-contrast and contrast echocardiography. These will be compared for identification of thrombi and assessment of cardiac size and function. Clinical features and results of other diagnostic tests will also be reviewed in order to study whether these predict thrombus risk. Participants will be contacted at regular intervals by study investigators to determine whether thrombi identified by contrast or non-contrast echocardiography predict risk for stroke or cardiac events. Findings from this study may improve detection of thrombi, thereby improving treatment for patients following myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* all patients who are admitted to The New York Presbyterian Hospital-Weill Medical College of Cornell University (NYP-WMC) with ST elevation myocardial infarctions

Exclusion Criteria:

* contraindications to MRI at time of planned imaging (e.g. metallic contra-indication, pacemaker, implantable cardiac defibrillator, cochlear implants, aneurysm clips intolerance of the imaging protocol due to NYHA IV heart failure or CCS class IV angina)
* known allergy/contra-indications to gadolinium or echo contrast agents (i.e. known intracardiac shunt, severe reactive airway disease)
* known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cross-sectional population of subjects enrolled following ST-elevation myocardial infarction.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2007-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan W Weinsaft, MD, Principal Investigator — Weill Medical College of Cornell University; Richard B Devereux, MD, Study Chair — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States

REFERENCES:
- [Derived] Weinsaft JW, Kim J, Medicherla CB, Ma CL, Codella NC, Kukar N, Alaref S, Kim RJ, Devereux RB. Echocardiographic Algorithm for Post-Myocardial Infarction LV Thrombus: A Gatekeeper for Thrombus Evaluation by Delayed Enhancement CMR. JACC Cardiovasc Imaging. 2016 May;9(5):505-15. doi: 10.1016/j.jcmg.2015.06.017. Epub 2015 Oct 14. PMID 26476503
- [Derived] Weinsaft JW, Kochav JD, Afroz A, Okin PM. Q wave area for stratification of global left ventricular infarct size: comparison to conventional ECG assessment using Selvester QRS-score. Coron Artery Dis. 2014 Mar;25(2):138-44. doi: 10.1097/MCA.0000000000000062. PMID 24300167
- [Derived] Chinitz JS, Chen D, Goyal P, Wilson S, Islam F, Nguyen T, Wang Y, Hurtado-Rua S, Simprini L, Cham M, Levine RA, Devereux RB, Weinsaft JW. Mitral apparatus assessment by delayed enhancement CMR: relative impact of infarct distribution on mitral regurgitation. JACC Cardiovasc Imaging. 2013 Feb;6(2):220-34. doi: 10.1016/j.jcmg.2012.08.016. PMID 23489536